CLINICAL TRIAL: NCT06744257
Title: Is Online Patient EducatioN Feasible in People With Patellofemoral Pain Whilst They Wait for Physiotherapy
Acronym: OPEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Suffolk and North Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21/228
Record Dates: First submitted 2024-11-22; First posted 2024-12-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Patello Femoral Syndrome
Keywords: Knee pain; Physiotherapy; Patellofemoral knee pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The Prinicipal Investigator of the study will be blinded to all individual participant information and only have access to unique pseudonymised study numbers/ data and which group they are assigned too.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online exercise program (Experimental): The online education arm will be provided with password access to our online patient education platform (https://www.teampfp.com/my-knee-cap-pain) that contains four modules; [a] Understand your pain; [b] How do I start to exercise; [c] Treatment options; [d] Case studies. The aim of each module is to provide people with knowledge they can put into practice (experiential learning) and facilitating their self-management. A short quiz at the end of each module assesses user engagement and knowledge retention.
  Interventions: Other: Online Education tool
- Standard of Care (No Intervention): The control arm will receive no additional care whilst on the ESNEFT physiotherapy waiting list. Their involvement in the trial will end at six-weeks follow up and they will then be provided with access to the online education platform if they request it.

INTERVENTIONS:
Other: Online Education tool — An online education tool that contains 4 modules
  Arms: Online exercise program

SUMMARY:
The primary aim is to determine if online patient education is a feasible intervention for people with PFP awaiting physiotherapy. The secondary aim is to provide outcome data to inform a future substantiative trial.

DETAILED DESCRIPTION:
Participants will take part in a feasibility trial whilst they are on the ESNEFT physiotherapy waiting list to avoid disrupting their routine care.

Participants will first attend a face-to-face eligibility assessment to validate their diagnosis of PFP, before being randomised to one of two arms:

1. The online education arm will be provided with password access to our online patient education platform (https://www.teampfp.com/my-knee-cap-pain) that contains four modules; [a] Understand your pain; [b] How do I start to exercise; [c] Treatment options; [d] Case studies. The aim of each module is to provide people with knowledge they can put into practice (experiential learning) and facilitating their self-management. A short quiz at the end of each module assesses user engagement and knowledge retention.

   Investigators developed these modules alongside members of the International Patellofemoral Research Network, and people with PFP that attended a PPI event at Queen Mary University London (QMUL) that aimed to understand what information people with PFP wanted to help them self-manage their condition.

   Participants randomised to the online education group will be instructed to consume the content at their own pace (with one module/week advised) and that their adherence will be determined by monitoring their completion of each end of module quiz. Participants with no access to a device or the internet, will be given a paper version.
2. The control arm will receive no additional care whilst on the ESNEFT physiotherapy waiting list. Their involvement in the trial will end at six-weeks follow up and they will then be provided with access to the online education platform if they request it.

The feasibility outcomes, adapted from those used in recent trials and mapped to trial quality appraisal scales, are designed to inform us on the willingness of clinicians to recruit participants, the willingness of participants to be randomised, if participants will accept and adhere to patient education intervention, if sufficient data can be collected, and potential effects of online education. Outcomes informing intervention effects have been optimised after discussion with participants from two pre-trial PPI focus groups. Outcome measures will be collected using the good data protection regulations (GDPR) compliant REDCap system (https://www.project-redcap.org/). Participants will receive regular prompts and paper versions with stamped/addressed envelopes will be available to those who are digitally illiterate, supported by a research assistant.

1. Recruitment and eligibility; a recruitment rate of four eligible participants per month is targeted, with consent rate (eligible/consenting participants) calculated
2. Randomisation and blinding; broad equality of baseline characteristics between groups and acceptable outcome assessor blinding will be targeted
3. Adherence and acceptability; >75% of participants in the online education arm attempting the end of education module quizzes and acceptability meaningfully greater than remaining on a waiting list
4. A maximum 20% attrition rate in either arm
5. Data collection; with >85% of participants completing all outcome measures at six-week follow up targeted.
6. The 7-point Likert global rating of change (GROC) scale will be used to allow comparison to recent RCTs involving people with PFP. Categories will be: [1] much better, [2] better, [3] a little better, [4] no change, [5] a little worse [6] much worse, and [7] markedly worse. Successful outcome will be dichotomised and defined a priori as [1] much better or [2] better at six-weeks follow up.
7. An eleven-point numerical pain rating scale (NPRS) will assess worst pain in the past week, which is valid and responsive in people with PFP 9.
8. The reliable and responsive EQ-5D-5L will assess health-related quality of life; important for future cost-effectiveness analyses 16. The final question of EQ-5D-5L relates to anxiety/depression. If participants select severely or extremely anxious or depressed, the investigators will inform the participant's GP.

Investigators will invite a subset of participants randomised to the online education arm to participate in a maximum of two semi-structured focus groups (n=6 per group) or 1:1 interviews post-trial. The aim of these focus groups will be to explore their perspectives on participating in our feasibility trial and receiving our online patient education intervention. Investigators will specifically explore the factors that affected if participants felt they had benefitted from receiving online patient education, and whether further physiotherapy input was still required. These semi-structured focus groups will be conducted by co-applicant Dr Katharine Fowler.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-44 years
* Gradual onset retro-and/or peri-patellar pain
* Symptoms reproduced during one or more of running; jumping; stair ambulation; squatting
* Referred to East Suffolk and North Essex NHS Foundation Trust for outpatient physiotherapy at Colchester hospital
* Able to read and understand written/spoken English

Exclusion Criteria:

* Aged 45 years and older
* Symptoms of concomitant knee pathology
* Symptoms commencing after trauma or knee surgery
* Presentation inconsistent with patellofemoral pain during clinical examination
* Unable to understand written/spoken English
* Unable to give informed consent

Ages: 16 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment and eligbility | From recruitment until end of follow up at 6 weeks.
  A recruitment rate of four eligible participants per month is targeted, with consent rate (eligible/consenting participants) calculated.
7-point likert scale | From recruitment until end of follow up at 6 weeks.
  We will use the 7-point Likert global rating of change (GROC) scale with categories: [1] much better, [2] better, [3] a little better, [4] no change, [5] a little worse [6] much worse, and [7] markedly worse. Successful outcome will be dichotomised and defined a priori as [1] much better or [2] better.
Adherence and acceptability rate | From recruitment until end of follow-up at 6 weeks
  >75% of participants in the online education arm attempting the end of education module quizzes and acceptability meaningfully greater than remaining on a waiting list.
Attrition rate | From recruitment until end of follow-up at 6 weeks
  A maximum 20% attrition rate in either arm.
Data collection | From recruitment until end of follow up at 6 weeks
  With >85% of participants completing all outcome measures at six-week follow up targeted.
NPRS scoring | From recruitment until end of follow up at 6 weeks.
  An eleven-point numerical pain rating scale (NPRS) will assess worst pain in the past week.
EQ-5D-5L (EuroQol Group-5 dimensions-5 levels) | From recruitment until end of follow up at 6 weeks.
  The reliable and responsive EQ-5D-5L will assess health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- East Suffolk and North Essex NHS Foundation Trust, Colchester, United Kingdom